CLINICAL TRIAL: NCT06037499
Title: Leistungsbewertungsprüfung Der Systemgenauigkeit, Von 14 Blutglukose Monitoring Systemen in Anlehnung an ISO 15197:2015
Brief Title: System Accuracy of 14 Blood Glucose Monitoring Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut fur Diabetes Karlsburg GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023_001
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subject glucometer measurement (Experimental)
  Interventions: Diagnostic Test: Glucometer Test

INTERVENTIONS:
Diagnostic Test: Glucometer Test — measurement of blood glucose concentration using different BGM and Reference Method

SUMMARY:
The system accuracy of 14 blood glucose monitoring systems is to be evaluated randomly in accordance with DIN EN ISO 15197:2015 over thr courese of 24 months

ELIGIBILITY:
Inclusion criteria:

* Male or female patients with hypo-, eu- or hyperglycaemia
* The written informed consent had to be signed
* The volunteers must be older than 18 years
* The volunteers have legal capacity and are able to understand meaning, nature and possible consequences of the procedures involved

Exclusion criteria:

* Pregnancy or lactation
* Acute or chronic diseases with the risk of aggravation by the measure
* A current constitution that does not allow participating in the study
* Participation in another study or activity with the blood glucose measuring system evaluated in the present study
* Application of substances listed in Appendix A of DIN EN ISO 15197:2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose measurement using BGMS | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes Karlsburg GmbH, Karlsburg, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No